CLINICAL TRIAL: NCT01214174
Title: A Multicenter, Randomized, Double-masked, Dose-ranging, Phase 2 Study to Evaluate the Efficacy and Safety of IBI-10090 in Treating Inflammation in Cataract Surgery Patients
Brief Title: Efficacy and Safety Study of IBI-10090 in Cataract Surgery Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study C11-01 started
Sponsor: ICON Bioscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C10-01
Record Dates: First submitted 2010-09-21; First posted 2010-10-04 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Ocular Inflammation
Keywords: cataract; inflammation
MeSH Terms: conditions — Cataract; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 (Experimental): 513ug
  Interventions: Drug: IBI-10090
- Dose 2 (Experimental): 776ug
  Interventions: Drug: IBI-10090
- Dose 3 (Experimental): 1046ug
  Interventions: Drug: IBI-10090

INTERVENTIONS:
Drug: IBI-10090

SUMMARY:
This study will test the efficacy and safety of IBI-10090 in the treatment of ocular inflammation after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 40 years of age scheduled for unilateral cataract surgery (phacoemulsification or extracapsular extraction) with posterior chamber intraocular lens implantation.

Exclusion Criteria:

* Patients who have used any ocular, topical, or oral corticosteroids within 7 days prior to Day 0.
* Patients who have used topical ocular NSAIDs in the study eye within 15 days prior to screening.
* Patients with any signs of intraocular inflammation in either eye at screening.
* Patients who have received any prior intravitreal injections in the study eye.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, Principal Investigator — Drs. Fine, Hoffman, Packer
Locations (1):
- Drs. Fine, Hoffman, and Packer, Eugene, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose 1: IBI-10090 513ug
- Dose 2: IBI-10090 776ug
- Dose 3: IBI-10090 1046ug
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3
Started | 13 | 16 | 14
Completed | 13 | 16 | 13
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Total
Number analyzed (Participants) | 13 | 16 | 13 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 7
  >=65 years | 11 | 13 | 11 | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 70.9 (5.5) | 72.4 (8.9) | 73.5 (7.2) | 72.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 17
  Male | 9 | 10 | 6 | 25
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Anterior Chamber Cell Clearing at Day 8 Post-Treatment
Description: This study will measure as its primary endpoint the anterior chamber cell count at Day 8 post-treatment in the study eye. The proportion of patients with anterior chamber cell count = 0 at Day 8 in the study eye for each dosage group will be compared. Only one eye was treated per participant.
Time Frame: 8 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with ACC clearing
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 13 | 16 | 13
percentage of patients with ACC clearing | 30.8 [5.68 to 55.86] | 25 [3.78 to 46.22] | 46.2 [19.05 to 73.25]

ADVERSE EVENTS:
Arm/Group | Dose 1 | Dose 2 | Dose 3
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/16 | 3/13
Other Adverse Events (participants affected / at risk) | 10/13 | 13/16 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=13) | Dose 2 (N=16) | Dose 3 (N=13)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Endophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=13) | Dose 2 (N=16) | Dose 3 (N=13)
Eye Disorders (Eye disorders) | 10 (13) | 13 (25) | 12 (19)
Infections and Infestations (Infections and infestations) | 1 (1) | 0 (0) | 5 (5)
Investigations (Investigations) | 2 (2) | 1 (1) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information related to this study is considered confidential information belonging to Icon Bioscience, Inc. Data on the use of the study drug and results of all clinical and laboratory studies are considered private and confidential. None of the details, results, or other information for this study shall be published or made known to a third party without written consent from Icon Bioscience, Inc., except for disclosure to regulatory agencies if required by law.